CLINICAL TRIAL: NCT00303082
Title: Clinical Trial for the Prevention of Premature Birth and Neonatal Related Morbidity
Brief Title: Probiotics for the Prevention of Premature Birth and Neonatal Related Morbidity
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Limitation of funding
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Leticia Krauss Silva, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MDTP2/PDTSP-SUS
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2009-10

CONDITIONS: Bacterial Vaginosis; Premature Birth; Sepsis; Periventricular Leukomalacia; Bronchopulmonary Dysplasia
Keywords: Probiotics; Bacterial Vaginosis; Premature birth; Intra-uterine Infection; Periventricular leukomalacia
MeSH Terms: conditions — Vaginosis, Bacterial; Premature Birth; Sepsis; Leukomalacia, Periventricular; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lactobacillus rhamnosus GR1 and Lactobacillus reuteri RC-14

SUMMARY:
The trial intends to evaluate the efficacy of specially designed probiotics to prevent premature birth and related neonatal morbidity associated to intra-uterine infection. The tested probiotics are efficacious to decrease the prevalence of bacterial vaginosis. The study hypothesis is that the early administration of those probiotics to pregnant women with bacterial vaginosis can prevent premature birth through antibiotic activity and modulation of the immune response to infection.

DETAILED DESCRIPTION:
The study is designed to be a randomized placebo-controlled double-blind trial that will screen asymptomatic low risk pregnant women without indication of elective premature birth admitted before the 20th week of pregnancy (Date of LMP and ultrasound) in prenatal care public services involved in the project in the city of Rio de Janeiro. Relevant prognostic factors will be registered: history of premature birth, race and low body index.

After clinical screening will be followed by a further screening process:

1. vaginal pH exam will be determined by taking a swab and rolling it on a glass slide that will be touched by a pH stick . This procedure will immediately exclude patients with pH < 4,5 from the next step;
2. The slides from patients with a vaginal pH > 4.4, will be Gram stained and interpreted according to the criteria of Nugent et al in order to select patients with BV or intermediate Nugent score (4-10). Patients with Nugent score below 4 will be excluded.

Pregnant women who are excluded from any of the above steps will be reassessed every 4 weeks, for new cases of BV/Intermediate score, during the next prenatal care visits, until they reach the 19th week.

BV/Intermediate patients will be randomized (centralized blocked randomization process), after signed informed consent, to receive either probiotics or placebo capsules twice a day (each capsule with probiotics shall contain > 1 million bacilli of each of 2 selected strains of lactobacillus: Lactobacillus rhamnosus GR1 and Lactobacillus reuteri RC-14).

Women shall take the capsules until they reach approximately the 24th week of gestation, the minimum duration of the treatment being 6 weeks (for those women randomized to the trial by the 20th week). Capsules will be maintained in refrigerators throughout the trial.

Pregnant women will receive the usual prenatal care at their institutions, which should follow the related evidence-based municipal guidelines.

Vaginal pH and Nugent scores will be assessed after the end of the treatment for both treatment groups, so to assess changes in those parameters as partial results regarding the efficacy of the study probiotics.

Randomized patients, whether compliant with the treatment regimens or not, will be followed up for the assessment of the trial endpoints: spontaneous premature birth (<37, <35, <32 weeks of pregnancy) and related neonatal events: early sepsis, bronchopulmonary dysplasia, periventricular leukomalacia and necrotizing enterocolitis, besides death and average hospital stay. Study personnel will abstract that information from delivery and neonatal records using a pre-tested questionnaire. Definitions and diagnostic methods used for identifying such conditions will be similar to those recommended by the Vermont- Oxford Network, issued in 2002.

The occurrence of adverse events will be monitored with a specific questionnaire.

The adherence to the treatment will be assessed with specific questioning of the pregnant woman and by counting the capsules contained in the bottles returned by them at each prenatal care visit. Reasons for non adherence, including the occurrence of adverse events, will be looked into in order to propitiate adherence whenever possible.

Special attention will be devoted to avoid undesirable psychological effects derived from the eventual labeling of women as high risk for premature birth.

Procedures to assure the concealment of the randomization and the blinding of the pregnant women (identical placebo) and study personnel, including caretakers and the technician who will be performing the pH and Nugent exams, are described in the protocol.

In order to add further explanatory power to the present trial, regarding the mechanisms of action of the study probiotics, a nested case-control study (1 case and 3 controls) will be carried out to determine the level of selected cytokines (IL-1B, IL1-ra and IL-6) at the vaginal fluid, before and after treatment, and the occurrence of TNF an IL 6(308 and 174) polymorphisms, and their association, individually and in interaction, with the study endpoints (cases). Special vaginal swabs (cytokines) and oral samples (polymorphisms) will be collected for those purposes and processed accordingly. Written informed consent will be also sought for such procedures.

The trial was approved by an Institutional Review Board which has sent it for final approval by the National Review Board.

************************************************************

Sample size to show efficacy of study probiotics for preventing premature birth less than 35 and 32 weeks (significance level of 0.05 and power of 0.80):

_____________________________________________________________________

Considering:

* that using the pH <4.5 as a cutoff point for the Nugent assessment will result in excluding around 40% of the clinically pre-selected women (Hauth et al,2003) but will only exclude a small percentage of women with Nugent´s Intermediate score and related preterm births,
* a non-adherence rate to the treatment regimens of about 5%,
* that the incidence in the placebo group of premature birth less than 35 weeks will be around 6%;
* and an efficacy rate of 50% for the study main end-point (premature birth),

the number estimated to be necessary for the randomization phase of the present trial, is about 1500 women.

To assess efficacy regarding premature birth less than 32 weeks, same significance level and power, the corresponding number is nearly 3000.

ELIGIBILITY:
Inclusion Criteria:

-Asymptomatic pregnant women with no indication of elective preterm delivery, before the 20th week of pregnancy

Exclusion Criteria:

* major malformations in present pregnancy
* cervical cerclage
* symptomatic vaginosis
* insulin dependent diabetes
* arterial hypertension
* Multiple gestation
* Antibiotic therapy in present pregnancy
* Syphilis or gonorrhea in present pregnancy
* asthma requiring chronic or intermittent therapy
* corticotherapy(recent or chronic)
* perinatal hemolytic disease
* Systemic Erit. Lupus

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Spontaneous premature birth (<37, <35, <32 weeks of pregnancy) | 24 weeks

SECONDARY OUTCOMES:
and related neonatal events: early sepsis, bronchopulmonary dysplasia, cystic periventricular leukomalacia, ventricular hemorrhage and retinopathy, besides neonatal death. | 28 weeks
Variation in Nugent Score (before/after intervention) | 9 weeks
Variation in selected cytokine levels(before/after intervention) | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Krauss-Silva, MD, Ph.D, Principal Investigator — Oswaldo Cruz Foundation
Locations (2):
- Brazil (2):
  - Hospital Maternidade Alexander Fleming, Rio de Janeiro, Rio de Janeiro
  - Hospital Maternidade Carmela Dutra, Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Background] Andrews WW. Cervicovaginal cytokines, vaginal infection, and preterm birth. Am J Obstet Gynecol. 2004 May;190(5):1179. doi: 10.1016/j.ajog.2004.04.016. No abstract available. PMID 15167814
- [Derived] Krauss-Silva L, Moreira ME, Alves MB, Braga A, Camacho KG, Batista MR, Almada-Horta A, Rebello MR, Guerra F. A randomised controlled trial of probiotics for the prevention of spontaneous preterm delivery associated with bacterial vaginosis: preliminary results. Trials. 2011 Nov 8;12:239. doi: 10.1186/1745-6215-12-239. PMID 22059409
- [Derived] Krauss-Silva L, Moreira ME, Alves MB, Rezende MR, Braga A, Camacho KG, Batista MR, Savastano C, Almada-Horta A, Guerra F. Randomized controlled trial of probiotics for the prevention of spontaneous preterm delivery associated with intrauterine infection: study protocol. Reprod Health. 2010 Jun 30;7:14. doi: 10.1186/1742-4755-7-14. PMID 20591191